CLINICAL TRIAL: NCT04343508
Title: Study to Evaluate the Efficacy of Fortified Rice on Hemoglobin Levels and Levels of Vitamins and Minerals in Healthy Asian Migrant Workers in Singapore
Brief Title: Impact of Fortified Rice on Workers' Nutrition Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Collaborators: Sprim Advanced Life Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OBVO-0104DSM
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Nutrient Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fortified rice (Experimental): fortified rice for daily lunch and dinner each day of the week (i.e. 14 meals/week) for six months
  Interventions: Other: Fortified rice

INTERVENTIONS:
Other: Fortified rice — 100 g of rice was fortified with 150 µg vitamin A (Vitamin A palmitate), 0.5 mg vitamin B1 (thiamin mononitrate), 7 mg vitamin B3 (niacin amide), 0.6 mg vitamin B6 (pyrodoxine hydrochloride), 1 µg vitamin B12 (cyanocobalamin), 130 µg folic acid, 4 mg iron (ferric pyrosphosphate), and 6 mg zinc (zinc oxide).

SUMMARY:
The study is a single center, open label, nutrition intervention study. Healthy adult male working at a Singapore construction site are included if they fulfill inclusion and exclusion criteria. Volunteers receive fortified rice for their daily lunch and dinner each day of the week (i e 14 meals/week) over six months. Nutrition status in blood is measured at baseline and after six months of fortified rice consumption.

DETAILED DESCRIPTION:
The study is a single center, open label, uncontrolled longitudinal nutrition intervention study. Migrant construction workers of either Bangladeshi or Indian ethnicity from a single dormitory in Singapore volunteer to participate at the study. Only eligible workers are included in the study if they fulfilled all inclusion and exclusion criteria; 20 and 51 years old, a BMI between 17.0 to 27.5 kg/m2, willing to adhere to the study procedure for at least six months, and sign informed consent, are free of current medical and/or chronic/non communicable diseases, no history of heavy smoking or alcohol consumption. The eligible subjects receive fortified rice for their daily lunch and dinner each day of the week (i e 14 meals/week) over six months. The nutrient levels per 100 g fortified rice contain 150 µg vitamin A (Vitamin A palmitate), 0.5 mg vitamin B1 (thiamin mononitrate), 7 mg vitamin B3 (niacin amide), 0.6 mg vitamin B6 (pyridoxine hydrochloride), 1 µg vitamin B12 (cyanocobalamin), 130 µg folic acid, 4 mg iron (ferric pyrosphosphate), and 6 mg zinc (zinc oxide). At baseline and after 6 months of intervention, BMI and vital signs such as blood pressure, pulse and body temperature are collected. Also, 10 ml venous blood is sampled at baseline and after 6 months of intervention and subsequently tested for hemoglobin, serum folate, and serum zinc, serum ferritin and serum vitamin B12 status. In a small subset of the migrant construction workers, an extra 5 ml blood sample is taken for homocysteine testing.

ELIGIBILITY:
Inclusion Criteria:

* 20 Years to 51 Years
* Indian or Bangladeshi ethnic origin
* BMI of 17.0 to 27.5 kg/m2
* Working at the construction site and continuing for 6 months after enrollment
* Willing and able to adhere to study procedures
* Signed the informed consent form

Exclusion Criteria:

* Conditions or diseases that the investigator considers to be not appropriate to enter the study
* Chronic illness
* History of heavy smoking (more than 10 cigarettes/day continuously for two years or more (self-reported) )
* Unable to understand informed consent (translated to Tamil and Bangladesh at basic literacy level)

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2018-03-11 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Hemoglobin status | From baseline to 6 months
  Hemoglobin concentration in blood

SECONDARY OUTCOMES:
Folate status | From baseline to 6 months
  Red blood cell folate concentration in serum
Zinc status | From baseline to 6 months
  Serum zinc concentration
Iron status | From baseline to 6 months
  Serum ferritin concentration
Vitamin B12 status | From baseline to 6 months
  Serum vitamin B12 concentration
Homocysteine status | From baseline to 6 months
  Serum homocysteine concentration
BMI | From baseline to 6 months
  BMI calculated from height and weight

OTHER OUTCOMES:
Height | From baseline to 6 months
  Height (cm)
Weight | From baseline to 6 months
  Weight (kg)
Blood pressure | From baseline to 6 months
  Systolic and Diastolic Blood Pressure (mmHg)
Pulse | From baseline to 6 months
  Pulse (count/min)
Body temperature | From baseline to 6 months
  Body temperature (degrees Celsius)

CONTACTS AND LOCATIONS:
Locations (1):
- SPRIM, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided